CLINICAL TRIAL: NCT06091345
Title: Midodrine Plus Albumin Versus Midodrine Alone to Prevent Cirrhosis Related Complications in Children With Cirrhosis and Ascites - An Open Label Randomized Controlled Trial.
Brief Title: Midodrine Plus Albumin Versus Midodrine Alone to Prevent Cirrhosis Related Complications in Children With Cirrhosis and Ascites
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Liver and Biliary Sciences, India (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ILBS-Cirrhosis-65
Record Dates: First submitted 2023-10-13; First posted 2023-10-19 (Actual); Last update posted 2025-07-01 (Actual); Status verified 2025-06

CONDITIONS: Liver Cirrhosis
MeSH Terms: conditions — Liver Cirrhosis | interventions — Midodrine; Albumins

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Midodrine+Albumin+SMT (Experimental): * Albumin infusion 1g/kg/day (max 20g) every two weeks (if pre-infusion serum albumin is < 3.5 gm/dl Plus
  * Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% .
  In addition, standard medical therapy will be administered to patients in both the arms.
  Interventions: Drug: Midodrine; Biological: albumin; Other: Standard Medical Treatment
- Midodrine+SMT (Active Comparator): • Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10% In addition, standard medical therapy will be administered to patients in both the arms.
  Interventions: Drug: Midodrine; Other: Standard Medical Treatment

INTERVENTIONS:
Drug: Midodrine — • Midodrine starting at 0.25mg/kg/day in divided doses, increased to 0.5mg/kg/day after 7 days if MAP does not increase by >10%
Biological: albumin — • Albumin infusion 1g/kg/day (max 20g) every two weeks (if pre-infusion serum albumin is < 3.5 gm/dl
  Arms: Midodrine+Albumin+SMT
Other: Standard Medical Treatment — Standard Medical Treatment

SUMMARY:
Children with decompensated cirrhosis are more prone to develop various complications. The pathogenesis of cirrhotic complications (ascites, hyponatremia, acute kidney injury) includes release of vasodilatory molecules like nitric oxide, damage associated molecular pathogens (DAMPs) and pattern associated molecular pathogens (PAMPs) secondary to bacterial translocation, which causes splanchnic bed vasodilation resulting in activation of renin-angiotensin and aldosterone axis (RAAS) causing sodium and water retention and renal vasoconstriction.

The development of complications in these children may result in death or may preclude them from reaching upto liver transplantation.

Midodrine is an α1 adrenergic receptor agonist, which increases vascular tone causing rise in the blood pressure, thereby improving renal perfusion and causes RAAS deactivation. The effects of midodrine is documented in reduction of refractory ascites, hepatorenal syndrome and hyponatremia.

Albumin is a protien that works by both increasing the colloidal oncotic pressure and improving systemic circulation as well as by effecting the body with anti-inflammatory and antioxidant properties.

We have already demonstrated the safety and efficacy of midodrine as well as albumin in cirrhotic children. However, none of these drugs alone provided survival benefit to the patients. Hence, we have planned this study with the ojective to evaluate if combining these 2 drugs (midodrine and albumin) would further reduce the complications and improve the survival in decompensated cirrhotic children.

DETAILED DESCRIPTION:
Aim: To evaluate whether a combination of midodrine and intravenous albumin reduces complications of cirrhosis in decompensated (ascites) cirrhotic children as compared to midodrine alone.

Primary objective: To compare difference in composite incidence of complications of cirrhosis (Acute kidney injury, ascites, hyponatremia, hepatic encephalopathy) in patients receiving midodrine and albumin versus those receiving midodrine alone.

Secondary objectives:

1. To compare the rate of control of ascites by 6 months in the 2 groups
2. To compare the change in Mean arterial pressure (MAP) at 1 week, 2 weeks, 4 weeks, 3 months, and 6 months in the 2 groups
3. To compare the Plasma renin activity at baseline, 4 weeks, 3mo, 6mo in the 2 groups
4. Evaluate the change in serum sodium from baseline to 6 months in the 2 groups
5. To compare the Creatinine from baseline to 6 months in the 2 groups
6. To compare the Frequency of development of drug related adverse effects by 6 months
7. To compare the Transplant free survival in the 2 groups
8. To compare the Cytokines levels at baseline and 6 months in the 2 groups
9. To compare the presence of Minimal Hepatic encephalopathy in the 2 groups Study population :Children and Adolescents of age group upto 18 years with decompensated cirrhosis with clinical ascites, following up in the Pediatric Hepatology Department, ILBS will be prospectively included in this study after informed consent

   * Study design: Open-label Randomized Controlled Trial
   * Study period: 6 months weeks for each patient; The study will be conducted from the time of ethical approval to June 2025.

Sample size: In a pilot trial done at our center comparing midodrine and SMT the composite incidence of complication was 61.2% in midodrine arm. In absence of a pediatric study we assume a 25% reduction of complication by adding albumin along with midodrine keeping a power of study 80% , the sample size was calculated to be 30 in each arm.

ELIGIBILITY:
Inclusion Criteria:

1. Children (≤ 18 years)
2. Cirrhosis based on histological/ radiological + endoscopic evidence
3. Clinical ascites (≥ grade 2 ascites)
4. Informed consent from parents (Assent > 12 years)

Exclusion Criteria:

1. Arterial hypertension (Mean Arterial Pressure ≥ 95th centile for age)
2. Presence of Portal vein thrombosis
3. Hepatorenal Syndrome
4. Congestive Heart failure
5. Respiratory failure(PF ratio <200)
6. Septic shock
7. Presence of Hepatocellular Carcinoma
8. Transjugular intrahepatic Porto Systemic Shunt

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 60 (Estimated)
Dates: Start 2023-11-02 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
To compare difference in composite incidence of complications of cirrhosis (Acute kidney injury, ascites, hyponatremia, hepatic encephalopathy) in patients receiving midodrine and albumin versus those receiving midodrine alone. | 6 months

SECONDARY OUTCOMES:
To compare the rate of control of ascites by 6 months in the 2 groups | 6 months
To compare the change in Mean arterial pressure (MAP) at 1 week, 2 weeks, 4 weeks, 3 months, and 6 months in the 2 groups | 1 week, 2 weeks, 4 weeks, 3 months, and 6 months
To compare the Plasma renin activity at baseline, 4 weeks, 3mo, 6mo in the 2 groups | baseline, 4 weeks, 3months, 6months
Evaluate the change in serum sodium from baseline to 6 months in the 2 groups | 6 months
To compare the Creatinine from baseline to 6 months in the 2 groups | 6 months
To compare the Frequency of development of drug related adverse effects by 6 months | 6 months
To compare the Transplant free survival in the 2 groups | 6 months
To compare the Cytokines levels at baseline and 6 months in the 2 groups | 6 months
To compare the presence of Minimal Hepatic encephalopathy in the 2 groups | 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Liver & Biliary Sciences (ILBS), New Delhi, National Capital Territory of Delhi, India

IPD SHARING:
Plan to Share IPD: No